CLINICAL TRIAL: NCT05713708
Title: Multicenter Registry for S-ICD Electrodes
Brief Title: S-ICD Electrode Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Other Study IDs: SICDLEAD
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: ICD Malfunction; Sudden Cardiac Death
Keywords: subcutaneous cardioverter-defibrillator; S-ICD; electrode malfunction; lead failure; battery depletion
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The subcutaneous implantable cardioverter defibrillator (S-ICD) is established in the prevention of sudden cardiac death, but recently a defect of the electrode's Sense-B component was reported in some patients. This lead to inadequate shocks due to noise. The cause and incidence of this defect are unknown. The manufacturer issued a warning regarding this defect and a possible premature depletion of the battery in some device. Independent data on the incidence of these issues is limited. Further data is needed to better understand the risk of these complications.

DETAILED DESCRIPTION:
The S-ICD therapy is an established treatment for primary and secondary prevention of sudden cardiac death. Recently, a report was published about a previously described complication of the electrode, in which a defect of the so-called Sense-B component is reported in a few affected patients. The defect of this component of the electrode leads to electrode noise and subsequent inadequate shocks. The cause of the defect and the incidence are currently unknown. The manufacturer Boston Scientific has issued a warning and advisory.

In addition to this advisory regarding the electrode of the S-ICD, there is also an active warning from the manufacturer regarding the possible premature exhaustion of the S-ICD battery. This is caused by an error in the manufacturing process of approximately 40,000 devices produced in 2018. The manufacturer estimates the incidence of premature battery exhaustion to be 4-15% within 5 years. Independent data on the incidence of premature exhaustion of these devices were initially scarce. The investigators conducted a retrospective data query in 2021 to capture the incidence of battery exhaustion at that time. The incidence was 3.7% after 5 years. The average follow-up time was only 3 years. The incidence of premature exhaustion increased significantly after 3 years, so data with a longer follow-up period is urgently needed.

Given that these data already show that the incidence of premature exhaustion increases significantly after 3 years and the observation period in the retrospective data was on average slightly under 3 years, a further query of the existing clinical data on the battery as part of this register is also planned. This would allow for a more accurate estimate of the risk of premature battery depletion.

ELIGIBILITY:
Inclusion Criteria:

- status post S-ICD insertion

Exclusion Criteria:

- no available follow-up data beyond 2 weeks after insertion

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received an S-ICD at the participating sites for whom meaningful follow-up data is available will be included.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-03 (Estimated)

PRIMARY OUTCOMES:
Sense B Electrode Failure | 3 months to 70 months after device insertion
  Incidence of the Sense B Electrode Failure of the S-ICD Lead.

SECONDARY OUTCOMES:
Premature Battery Depletion | 3 months to 70 months after device insertion
  Incidence of battery depletion of the S-ICD generator after insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luker J, Strik M, Andrade JG, Raymond-Paquin A, Elrefai MH, Roberts PR, Perez OC, Kron J, Koneru J, Franqui-Rivera H, Sultan A, Ernst A, Schmitt J, Pott A, Veltmann C, Srinivasan NT, Collinson J, van Stipdonk AMW, Linz D, Fluschnik N, Tonnis T, Haeberlin A, Ploux S, Steven D. Incidence of premature battery depletion in subcutaneous cardioverter-defibrillator patients: insights from a multicenter registry. J Interv Card Electrophysiol. 2025 Oct;68(7):1409-1415. doi: 10.1007/s10840-023-01468-1. Epub 2023 Jan 18. PMID 36652082
- [Background] Haeberlin A, Burri H, Schaer B, Koepfli P, Grebmer C, Breitenstein A, Reichlin T, Noti F. Sense-B-noise: an enigmatic cause for inappropriate shocks in subcutaneous implantable cardioverter defibrillators. Europace. 2023 Feb 16;25(2):767-774. doi: 10.1093/europace/euac202. PMID 36353759
- [Derived] Wormann J, Strik M, Jurisic S, Stout K, Elrefai M, Becher N, Schaer B, van Stipdonk A, Srinivasan NT, Ploux S, Breitenstein A, Kron J, Roberts PR, Toennis T, Linz D, Dulai R, Hermes-Laufer J, Koneru J, Erkuner O, Dittrich S, van den Bruck JH, Schipper JH, Sultan A, Rosenberger KD, Steven D, Luker J. Occurrence of premature battery depletion in a large multicentre registry of subcutaneous cardioverter-defibrillator patients. Europace. 2024 Jul 2;26(7):euae170. doi: 10.1093/europace/euae170. PMID 38885309
- [Derived] Wormann J, Strik M, Jurisic S, Stout K, Elrefai M, Becher N, Schaer B, van Stipdonk A, Srinivasan NT, Ploux S, Breitenstein A, Kron J, Roberts PR, Toennis T, Linz D, Dulai R, Hermes-Laufer J, Koneru J, Erkuner O, Dittrich S, van den Bruck JH, Schipper JH, Sultan A, Rosenberger KD, Steven D, Luker J. Incidence, implications, and management of sense-B-noise failure in subcutaneous cardioverter-defibrillator patients: insights from a large multicentre registry. Europace. 2024 Jun 3;26(6):euae161. doi: 10.1093/europace/euae161. PMID 38861398